CLINICAL TRIAL: NCT04455841
Title: A Phase 1/2 Open-Label, Multicenter Study of INCB000928 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Anemia Due to Myeloproliferative Disorders
Brief Title: INCB000928 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Anemia Due to Myeloproliferative Disorders
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 00928-104; 2023-503625-19-00 (Registry Identifier: EU CT Number); 2020-004029-21 (EudraCT Number)
Record Dates: First submitted 2020-06-19; First posted 2020-07-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Post-essential Thrombocythemia Myelofibrosis; Post-polycythemia Vera Myelofibrosis
Keywords: anemia
MeSH Terms: conditions — Anemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (TGA) (Experimental): INCB000928 will be administered once daily (QD).
  Interventions: Drug: INCB000928
- Treatment Group B (TGB) (Experimental): INCB000928 will be administered in combination with ruxolitinib.
  Interventions: Drug: INCB000928; Drug: ruxolitinib
- Treatment Group C (TGC) (Experimental): INCB000928 will be administered in combination with ruxolitinib.
  Interventions: Drug: INCB000928; Drug: ruxolitinib

INTERVENTIONS:
Drug: INCB000928 — INCB000928 will be administered at protocol defined dose.
Drug: ruxolitinib — Ruxolitinib will be administered at protocol defined dose.
  Arms: Treatment Group B (TGB); Treatment Group C (TGC)

SUMMARY:
This Phase 1/2, open-label, dose-finding study is intended to evaluate the safety and tolerability, PK, PD, and efficacy of INCB000928 administered as monotherapy or in combination with ruxolitinib in participants with MF who are transfusion-dependent or presenting with symptomatic anemia. This study will consist of 2 parts: dose escalation and expansion.

ELIGIBILITY:
Inclusion Criteria:

* Participants with MF who are transfusion-dependent or present with symptomatic anemia, defined as follows:

  1. Anemia: An Hgb value < 10 g/dL demonstrated during screening recorded on 3 separate occasions with at least 7 days between measurements (Note: RBC transfusion must be at least 2 weeks before the Hgb measurement during screening).
  2. Transfusion-dependent: Participant has received at least 4 units of RBC transfusions during the 28 days immediately preceding Cycle 1 Day 1 OR has received an average of at least 4 units of RBC transfusions in the 8 weeks immediately preceding Cycle 1 Day 1, for an Hgb level of < 8.5 g/dL, in the absence of bleeding or treatment-induced anemia. In addition, the most recent transfusion episode must have occurred in the 28 days before Cycle 1 Day 1.
* ECOG performance status score of the following:

  1. 0 or 1 for the dose-escalation stages.
  2. 0, 1, or 2 for the dose-expansion stage.
* Life expectancy is greater than 6 months
* Agreement to avoid pregnancy or fathering children.
* Ineligible to receive or have not responded to available therapies for anemia such as ESAs.
* For TGA:
* Participants previously treated with JAK inhibitors for at least 12 weeks.
* Participants with intermediate-2 or high DIPSS MF according to IWG-MRT criteria.
* For TGB:
* Participants must have been on a therapeutic and stable regimen of ruxolitinib for at least 12 consecutive weeks immediately preceding the first dose of study treatment.
* Participants with intermediate-1, intermediate-2, or high DIPSS MF according to IWG-MRT criteria.
* For TGC:
* Participants must be JAK inhibitor treatment naive (no prior treatment with any JAK inhibitor) and have an indication for initiation of ruxolitinib treatment.
* Participants with intermediate-1, intermediate-2, or high DIPSS MF according to IWG-MRT criteria.

Exclusion Criteria:

* Undergone any prior allogenic or autologous stem cell transplantation or a candidate for such transplantation.
* Any prior chemotherapy, immunomodulatory drug therapy, immunosuppressive therapy, biological therapy, endocrine therapy, targeted therapy, antibody or hypomethylating agent to treat the participant's disease, with the exception of ruxolitinib for TGB only, within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Laboratory Values outside of protocol defined range at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related adverse events | Approximately up to 13 months
  To determine the safety and tolerability of INCB000928 administered as monotherapy (TGA) or in combination with ruxolitinib (TGB and TGC).

SECONDARY OUTCOMES:
Anemia Response | Approximately up to 13 months
  Defined as an increase in hemoglobin.
Duration of Anemia Response | Approximately up to 13 months
  Duration of anemia response at baseline.
Mean Change of Hemoglobin | Approximately up to 13 months
  Mean change in hemoglobin levels from baseline.
Rate of RBC transfusion | Approximately up to 13 months
  Defined as the average number of RBC units.
TGB and TGC only -Splenic Volume | Approximately up to 13 months
  Defined as the proportion of participants achieving a targeted reduction in spleen volume.
TGB and TGC Only - Splenic Length | Approximately Up to 13 months
  Defined as the proportion of participants achieving a targeted reduction in spleen length.
TGB and TGC only - Objective Response Rate | Approximately up to 13 months
  Defined as the proportion of participants with Complete Response or Partial Response.
TGB and TGC only - Progression Free Survival | Approximately up to 13 months
  Defined as the interval from the first dose of study treatment until the first documented progression or death.
TGB and TGC only - Leukemia Free Survival | Approximately upto 13 months
  Defined as the interval from the first dose of study treatment until the first documented leukemia transformation or death from any cause.
AUC | Approximately up to 13 months
  Area Under the Plasma Concentration versus Time curve of INCB 00928-104.
Tmax | Approximately up to 13 months
  Time to reach maximum (peak) plasma concentration of INCB 00928-104.
AUC0-t | Approximately up to 13 months
  Area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t.
Hepcidin levels | Approximately up to 13 months
  Effect of INCB000928 administered as monotherapy (TGA) or in combination with ruxolitinib (TGB and TGC) on hepcidin levels.
Iron Homeostasis | Approximately up to 13 months
  Effect of INCB000928 administered as monotherapy (TGA) or in combination with ruxolitinib (TGB and TGC) on iron homeostasis parameters such as TSI, ferritin, transferrin, TSAT, TIBC, UIBC, and serum NTBI.
Erythropoesis | Approximately up to 13 months
  Effect of INCB000928 administered as monotherapy (TGA) or in combination with ruxolitinib (TGB and TGC) on erythropoiesis parameters such as RC, NRBC, MCV, MCH, Hgb, Hct, RBC count, MCHC, and RDW.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda McBride, MD, Study Director — Incyte Corporation
Locations (34):
- United States (13):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County, Irvine, California
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Prebys Cancer Center, San Diego, California
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - Start Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical Centers, New York, New York
  - Duke University Medical Center, Department of Hematologic Malignancies and Cellular Therapy, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Jewish General Hospital, Montreal, Quebec
- France (3):
  - Centre Hospitalier D'Angers, Angers
  - Institut Paoli Calmettes, Marseille
  - Hospital Saint Louis, Paris
- Italy (6):
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - S Orsolas University Hospital Seragnoli Institute of Hematology, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga Orbassano, Orbassano
  - Comitato Di Bioetica Della Fondazione Irccs Policlinico San Matteo, Pavia
  - Ospedale Santa Maria Della Misericordia Perugia, Perugia
- Japan (6):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Gifu Municipal Hospital, Gifu
  - Kansai Medical University Hospital, Hirakata
  - Kumamoto Shinto General Hospital, Kumamoto
  - Osaka International Cancer Institute, Osaka
- United Kingdom (4):
  - University Hospital of Wales, Cardiff, WLS
  - United Lincolnshire Hospitals, Boston
  - Lincoln County Hospital, Lincoln
  - Royal Cornwall Hospital Truro Sunrise Centre, Truro

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Related Info — https://www.incyteclinicaltrials.com/limber/